CLINICAL TRIAL: NCT05950880
Title: Effect of Adding High Intensity Exercises to Conventional Physical Therapy in Treatment of Athlete Patients With Shoulder Impingement Syndrome
Brief Title: Effect of High Intensity Exercises in Treatment of Patients With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdallah Gamiel Ayed, Mr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004361
Record Dates: First submitted 2023-07-05; First posted 2023-07-18 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity exercise + Conventional physical therapy (Experimental): Patients in this group will receive High-intensity exercise + Conventional physical therapy
  Interventions: Other: High intensity shoulder exercise; Other: Conventional physical therapy
- Conventional physical therapy (Active Comparator): Patients in this group will receive Conventional physical therapy
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: High intensity shoulder exercise — Exercises that target the rotator cuff muscles using 90% of one repetition maximum only for 5 repetitions
  Arms: High intensity exercise + Conventional physical therapy
Other: Conventional physical therapy — Conventional physical therapy consisting of scapular stabilization exercises, posterior capsule stretch, and rotator cuff activation exercises

SUMMARY:
Purposes of the study

To investigate the effect of adding High-Intensity Exercises to conventional physical therapy in patients with Shoulder Impingement Syndrome

DETAILED DESCRIPTION:
Patients will be randomized into either High-intensity shoulder exercise group or Conventional physical therapy group. Patients will receive the intervention for six weeks. Outcomes will be assessed at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Athletic patients
2. Age of the patients between 18 - 35 years
3. Unilateral shoulder pain more than 3 months.
4. Positive Hawkins test.
5. Positive empty or full cane test.
6. Pain at night or incapable of lying on the shoulder.
7. Pain with active shoulder elevation in the scapular plane.
8. History of pain in the C5-C6 dermatome.
9. Pain with palpation of the rotator cuff tendons.
10. The patient had pain with resisted isometric abduction

Exclusion Criteria:

1. History of shoulder instability (positive Sulcus sign, positive apprehension test, and history of shoulder dislocation).
2. Clinical sign of cervical radiculopathy.
3. History of acromio -clavicular pain.
4. Rheumatoid Arthritis.
5. Adhesive capsulitis.
6. Tumors
7. Labrum lesions
8. Capsular or ligamentous tears or avulsions
9. Cartilage lesions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
pain and function | Change from Baseline pain and function at 6 weaks
  Shoulder pain and disability index (SPADI)
Supraspinatus muscle thickness | Change from Baseline Supraspinatus muscle thickness at 6 weaks
  Diagnostic Ultrasound

SECONDARY OUTCOMES:
Sub acromial space (Acromiohumeral distance). | Change from Baseline Sub acromial space at 6 weaks
  Diagnostic Ultrasound
External and internal rotators muscle strength. | Change from Baseline External and internal rotators muscle strength at 6 weaks
  Hand-held dynamometer
supuraspinatus muscle strength | Change from Baseline supuraspinatus muscle strength at 6 weaks
  Hand-held dynamometer
shoulder performance | Change from Baseline shoulder performance at 6 weaks
  Timed push up test

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Gamiel, MSc, Principal Investigator — Cairo University
Locations (1):
- facult of physical therapy,MTI, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No